CLINICAL TRIAL: NCT05214547
Title: Focal Vibration Therapy Effectiveness in the Treatment of Patients With Adhesive Capsulitis
Brief Title: Effectiveness of Focal Vibration in Shoulder Pathology
Acronym: FVinAC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bitlis Eren University (Other)
Responsible Party: Principal Investigator, Tülay Çevik Saldıran, Associate Professor, Bitlis Eren University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BEU_FV
Record Dates: First submitted 2022-01-14; First posted 2022-01-28 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Adhesive Capsulitis; Shoulder
Keywords: Pain, Shoulder; Vibration
MeSH Terms: conditions — Bursitis; Shoulder Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Focal Vibration Group Training with Focal Vibration on the deltoid, trapezius, and biceps muscles with an amplitude of 1.2 mm. Time of training 20-25 min. The configuration of the vibration program will be in an automatic mode of 10 seconds of vibration and 3 seconds of rest to avoid the coupling of the mechanoreceptors. Patients will be treated with FV for three consecutive days: each session consisted of three sessions of 10 minutes each, interspersed with one minute of rest. A vibration frequency of 40 Hz to 100 Hz has been applied, according to the literature. The group also received the Traditional Training.
  Interventions: Device: Focal VibrationTherapy
- Control Group (Active Comparator): Traditional Training Warm up, grade 1 and 2 mobilization and stretching exercises, strength training, range of motion exercises, and coordination training.
  The home exercises program is programmed.
  Interventions: Device: Focal VibrationTherapy

INTERVENTIONS:
Device: Focal VibrationTherapy — Myovolt delivers oscillatory mechanical vibration of focussed frequency and low amplitude to stimulate physiological benefits in soft tissues. Myovolt is non-aggressive and gentle to the body so can be safely targeted. Digitally tuned to transmit a discrete vibration frequency range between 30 - 100Hz for effective neuromuscular stimulation.

SUMMARY:
We hypothesize that focal vibration therapy will reduce pain, increase the mobilization of the glenohumeral joint, and will improve functionality in patients with adhesive capsulitis.

DETAILED DESCRIPTION:
The underlying mechanism of focal vibration therapy in individuals with adhesive capsulitis still remains unclear. Considering the physiological mechanism of focal vibration therapy, the effect of focal vibration therapy on pain, function, and resting muscle tone in patients with adhesive capsulitis will be evaluated. There are no studies examining the effect of focal vibration therapy on shoulder muscle tone in individuals with adhesive capsulitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged > 18 years
* Unilateral adhesive capsulitis of the shoulder
* The symptom duration > 3 months
* Shoulder pain
* The limited glenohumeral joint active range of motion of greater than 50% in at least three specific movements among abduction, flexion, internal rotation, and external rotation

Exclusion Criteria:

* Previous shoulder surgeries
* Massive, minor, and major rotator cuff tears
* Pain and muscle strength loss due to neurological causes
* History or presence of malignancy
* Osteoporosis
* Diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-02-25 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-06-25 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Shoulder Pain at 4 weeks | At 4 week
  Evaluation of shoulder pain was performed using the Visual Analog Scale. The score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" on the far left and "the most intense pain imaginable" on the far right.The patient places a mark at a point on the line corresponding to the patient's rating of pain intensity. A higher score indicates greater pain intensity.
Change from 4 weeks Shoulder Pain at 6 weeks | At 6 week
  Evaluation of shoulder pain was performed using the Visual Analog Scale. The score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" on the far left and "the most intense pain imaginable" on the far right.The patient places a mark at a point on the line corresponding to the patient's rating of pain intensity. A higher score indicates greater pain intensity.

SECONDARY OUTCOMES:
Change from Baseline Range of Motion of Shoulder Joint at 4 weeks | At 4 weeks
  The joint movements of the affected shoulder was measured using a digital electrogoniometer. A higher score indicates greater improvement.
Change from 4 weeks Range of Motion of Shoulder Joint at 6 weeks | At 6 weeks
  The joint movements of the affected shoulder was measured using a digital electrogoniometer. A higher score indicates greater improvement.
Change from Baseline Shoulder Function at 4 weeks | At 4 weeks
  Function was assessed using the self-administered Shoulder Pain and Disability Index.The Shoulder Pain and Disability Index contains 13 items that assess two domains; a 5-item subscale that measures pain and an 8-item subscale that measures disability. Each subscale is summed and transformed to a score out of 100. A mean is taken of the two subscales to give a total score out of 100, higher score indicating greater impairment or disability.
Change from 4 weeks Shoulder Function at 6 weeks | At 6 weeks
  Function was assessed using the self-administered Shoulder Pain and Disability Index.The Shoulder Pain and Disability Index contains 13 items that assess two domains; a 5-item sub-scale that measures pain and an 8-item sub-scale that measures disability. Each sub-scale is summed and transformed to a score out of 100. A mean is taken of the two sub-scales to give a total score out of 100, higher score indicating greater impairment or disability.

OTHER OUTCOMES:
Change from baseline Shoulder Muscle Tone at 6 weeks | At 6 weeks
  The muscle tone which is a biomechanical property of the shoulder muscles will be evaluated with a portable hand-held myotonometer. This myotonometer (MyotonPRO - Tallinn, Estonia) is non-invasive and provides a quantitative assessment of a muscle's biomechanical properties. The MyotonPRO applies a short-intensity mechanical impulse on the skin overlying the muscle. The tissue's response then generates a signal that is recorded, and an internal software program produces an acceleration graph.

CONTACTS AND LOCATIONS:
Overall Officials: Tülay Çevik Saldıran, Ph.D., Study Director — Bitlis Eren University
Locations (1):
- Bitlis Eren University, Bitlis, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No